CLINICAL TRIAL: NCT05382156
Title: A Non-interventional Study to Assess the Long-term Safety and Efficacy of Osilodrostat in Patients With Endogenous Cushing's Syndrome
Brief Title: Non-interventional Study on Osilodrostat in Patients With Endogenous Cushing's Syndrome
Acronym: LINC6
Status: Active, not recruiting | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: LCI699-RECAG-PASS-0572
Record Dates: First submitted 2022-05-03; First posted 2022-05-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Endogenous Cushing's Syndrome
Keywords: Cushing's syndrome; Osilodrostat
MeSH Terms: conditions — Cushing Syndrome | interventions — Osilodrostat

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Osilodrostat: Osilodrostat - tablets of 1mg, 5mg, 10mg - based on patients needs - up to 3 years
  Interventions: Drug: Osilodrostat

INTERVENTIONS:
Drug: Osilodrostat — oral administration of Osilodrostat tablets at different doses according to patient's need
  Other Names: Isturisa

SUMMARY:
This is a non-interventional, multinational, multi-centre study with primary data collection, to further document the safety and efficacy of osilodrostat administered in routine clinical practice in patients treated with osilodrostat for endogenous Cushing's Syndrome

DETAILED DESCRIPTION:
This is a non-interventional, multinational, multi-centre study with primary data collection, to further document the safety and efficacy of osilodrostat administered in routine clinical practice in patients treated with osilodrostat for endogenous Cushing's Syndrome. This study is observational in nature and does not impose a therapy protocol, diagnostic/therapeutic interventions or a visit schedule.

Patients with endogenous Cushing's Syndrome who are treated with osilodrostat alone or in combination with other therapies will be considered eligible for study enrolment. Each patient enrolled in the study will be followed up for 3 years from study entry. Patients who discontinue prior to the end of the 3-year period will be followed-up for 3 months after discontinuation of osilodrostat and will be included in the analysis.

The total number of patients enrolled in this study will be approximately 201. Assuming a recruitment period of 3 years, the total study duration from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) will be 6 years. The maximum duration for the individual patient is 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to registration of any patient data
* Male or female patients aged 18 years or older with endogenous CS treated with osilodrostat. Treatment with osilodrostat can either be initiated at the first visit of the study or can have been initiated before screening.

Exclusion Criteria:

* Patients with exogenous CS
* Patients with Pseudo CS
* Patients participating in an interventional clinical trial with an investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will consist of adult male and female patients with endogenous Cushing's Syndrome. Eligible patients for the study must be treated with osilodrostat. Investigators need to ensure that patients enrolled in this study meet the study inclusion and exclusion criteria listed in the protocol.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of osilodrostat-related adverse events and serious adverse events | 3 years of treatment with osilodrostat
  Number of participants with Adverse Events and Serious Adverse Events

SECONDARY OUTCOMES:
Short and long-term efficacy of osilodrostat | at baseline before treatment start, after 1 month of treatment, then every 3 months in the first year and every 6 months thereafter through study completion up to three years
  Complete response rate: proportion of enrolled patients with mean Urinary Free Cortisol (mUFC) ≤ ULN
Short and long-term efficacy of osilodrostat | at baseline before treatment start, after 1 month of treatment, then every 3 months in the first year and every 6 months thereafter through study completion up to three years
  Partial response rate: proportion of enrolled patients with ≥ 50% reduction from baseline in mean urinary free cortisol (mUFC), (but mUFC > ULN)
Short and long-term efficacy of osilodrostat | at baseline before treatment start, after 1 month of treatment, then every 3 months in the first year and every 6 months thereafter through study completion up to three years
  Overall response rate: proportion of enrolled patients with mean urinary free cortisol (mUFC) ≤ ULN or at least 50% reduction from baseline
Changes in pituitary tumour size | at baseline before treatment start, after 6 months of treatment, then every 12 months through study completion up to three years
  Actual and percentage change from baseline in pituitary tumour size
Incidence of Adverse Events (Safety and Tolerability) | 3 years of treatment with osilodrostat
  Incidence of adverse events and laboratory abnormalities using the National Cancer Institute-Common Toxicology Criteria (NCI-CTC) grading scale (version 5.0).
Change of mean urinary free cortisol (mUFC) | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in mean urinary free cortisol (mUFC)
Change of Serum Cortisol | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in Serum Cortisol
Change of Late Salivary Cortisol | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in Late Salivary Cortisol
Change of adrenocorticotropic hormone (ACTH) | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in adrenocorticotropic hormone (ACTH)
Normalization of Serum Cortisol | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Proportion of patients achieving normalisation of Serum Cortisol
Normalization of Late Salivary Cortisol | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Proportion of patients achieving normalisation of Late Salivary Cortisol
Normalization of adrenocorticotropic hormone (ACTH) | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Proportion of patients achieving normalisation of adrenocorticotropic hormone (ACTH)
Change in Fasting Glucose | at baseline before treatment start, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in fasting glucose
Change in HbA1c | at baseline before treatment start, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in HbA1c
Change in Fasting Lipid Profile | at baseline before treatment start, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in Fasting Lipid Profile
Change in Serum Insulin | at baseline before treatment start, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in Serum Insulin
Change in Blood Pressure | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in Blood Pressure
Change in Body Weight | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in Body Weight
Change in Body Mass Index (BMI) | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in Body Mass Index (BMI)
Change in Waist Circumference | at baseline before treatment start, after 1 month of treatment, then every 3 months through study completion up to three years
  Actual and percentage change from baseline in Waist Circumference
Change in Facial Rubor | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Change from baseline in incidence and grade of severity at physical examination of the Cushing's syndrome clinical feature Facial Rubor
Change in Hirsutism | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Change from baseline in incidence and grade of severity at physical examination of the Cushing's syndrome clinical feature Hirsutism
Change in Striae | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Change from baseline in incidence and grade of severity at physical examination of the Cushing's syndrome clinical feature Striae
Change in Supraclavicular fat pad | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Change from baseline in incidence and grade of severity at physical examination of the Cushing's syndrome clinical feature Supraclavicular fat pad
Change in Dorsal fat pad | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Change from baseline in incidence and grade of severity at physical examination of the Cushing's syndrome clinical feature Dorsal fat pad
Change in Proximal muscle wasting (atrophy) | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Change from baseline in incidence and grade of severity at physical examination of the Cushing's syndrome clinical feature Proximal muscle wasting (atrophy)
Change in Central (abdominal) obesity | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Change from baseline in incidence and grade of severity at physical examination of the Cushing's syndrome clinical feature Central (abdominal) obesity
Change in Ecchymoses (bruises) | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Change from baseline in incidence and grade of severity at physical examination of the Cushing's syndrome clinical feature Ecchymoses (bruises)
Changes in Patient-Reported Outcome (PRO) questionnaire Cushing Quality of Life (QoL) | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Actual and percentage change from baseline in score of PRO questionnaire CushingQoL. The minimum and maximum values are 12 and 60 respectively, where higher score means a better outcome
Changes in Patient-Reported Outcome (PRO) questionnaire Euro Quality of Life (EQ) - 5 Dimensions (5D) - 5 Levels (5L) | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Actual and percentage change from baseline in score of PRO questionnaire EQ-5D-5L. The minimum and maximum values for the questions are 11111 and 55555 respectively, where higher score is a worst outcome. For the visual analogue scale minimum and maximum values are 0 and 100 respectively, where higher score means a better outcome
Changes in Patient-Reported Outcome (PRO) questionnaire Beck Depression Inventory II (BDI-II) | at baseline before treatment start, after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Actual and percentage change from baseline in score of PRO questionnaire BDI-II. The minimum and maximum values are 1 and 63 respectively, where higher score means a worse outcome
Changes in Patient-Reported Outcome (PRO) questionnaire Patient Global Impression of Change (PGIC) | after 3 months of treatment, after 6 months of treatment, then every 6 months through study completion up to three years
  Actual and percentage change in score of PRO questionnaire PGIC. The minimum and maximum values of the question are 1 and 7 respectively, where higher score means a better outcome. For the visual analogue scale minimum and maximum values are 0 and 10 respectively, where higher score means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mario Maldonado, MD, Study Chair — Recordati AG - Head of Clinical Development
Locations (43):
- United States (15):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Emory University School, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University Schl-med, Indianapolis, Indiana
  - St Elizabeth Physicians, Covington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Grossman School of Medicine, New York, New York
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - New York, New York, New York
  - Endocrinology Research Associates, Inc., Columbus, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Froedtert Hospital, Milwaukee, Wisconsin
- France (10):
  - Hôpital Haut-Lévêque, Bordeaux
  - Hospices Civiles de Lyon, Bron
  - CHU de Grenoble site Nord, Grenoble
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hopital Claude Huriez - CHRU Lille, Lille
  - Hopital de la Conception - APHM, Marseille
  - Hôpital de Brabois, Nancy
  - CHU de Nantes-Hopital Laennec, Nantes
  - Hôpital Cochin, Paris
  - Hopital Larrey, Toulouse
- Germany (11):
  - Charité Universitaetsmedizin Berlin, Berlin
  - Medicover Berlin-Mitte MVZ, Berlin
  - Medicover Köln, Cologne
  - Universitaet Bielefeld - Klinikum Bielefeld - Mitte, Düsseldorf
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt
  - Endokrinologikum Frankfurt, Frankfurt
  - Amedes Experts, Hamburg
  - Medicover Neuroendokrinologie, Munich
  - Ludwig-Maximilians University of Munich, Munich
  - Medicover MVZ Oldenburg, Oldenburg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Italy (5):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Ancona
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Policlinico Umberto I, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
- Netherlands (2):
  - Radboud University Nijmegen, Nijmegen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes